CLINICAL TRIAL: NCT01295203
Title: Internet-based Physical Activity Intervention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Andreas Wolff Hansen, National Institute of Public Health, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NIPH 1957
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2008-05

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Control group (No Intervention): The control group were not given access to the intervention website and received no additional information.
  Interventions: Behavioral: website assess

INTERVENTIONS:
Behavioral: website assess — The internet intervention group were given assess to the intervention website which included a personal page with tailored physical activity advice and a personal profile together with Recommendations and general training programs.

SUMMARY:
The purpose of this study is to determine whether access to a website with personalized feedback on physical activity level and suggestions to increase physical activity results in improvements in self-reported physical activity, anthropometrics and physiological measurements

DETAILED DESCRIPTION:
In a website-based intervention study, the investigators wish to examine if it is possible to increase physical activity among inactive persons. Main objective is to determine if access to a website with personalized feedback on PA level and suggestions to increase PA results in improvements in self reported PA, anthropometrics and applied physiological measurements.

Physical inactive adults (n=12,287) participating in a nationwide health survey and examination (DANHES) were asked to randomly assigned to either intervention (n=6,055) or control group (n=6,232). The intervention group had access to a PA website with personalized advice and suggestions to increase PA. After 3 and 6 months, a follow-up questionnaire was administered by e-mail. The 7-day International Physical Activity Questionnaire was included in the questionnaires to assess four domains of PA in daily-life (work, transportation, domestic, and leisure-time) and sedentary time. Furthermore, at the 3 month follow-up a subgroup of participants (n=1,190) were invited complete anthropometrics and physiological measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Physically inactive in leisure time (assessed by self reported questionnaire)

Exclusion Criteria:

* Presence of serious heart problems or not being able to perform everyday activities
* Highly physically active in leisure time (assessed by self reported questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12287 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Self reported physical activity | after 3 month
  Physical activity was assessed self reported with the International Physical Activity Questionnaire (IPAQ)
Self reported physical activity | After 6 month
  Physical activity was assessed self reported with the International Physical Activity Questionnaire (IPAQ)

SECONDARY OUTCOMES:
Body weight | after 3 month
  Body weight was measured to the nearest 0.1 kg and percent point with a Segmeantal Body Composition Analyser (type BC-418 MA, Tanita Corp., Tokyo, Japan).
Fat percentage | after 3 month
  Fat percentage was measured to the nearest 0.1 kg and percent point with a Segmeantal Body Composition Analyser (type BC-418 MA, Tanita Corp., Tokyo, Japan).
Hip and Waist circumference | after 3 month
  Hip and waist circumference was measured with a body tape (Chasmors WM02 Body Tape, Chasmors Ltd.,London, United Kingdom) to the nearest 1.0 cm. Waist circumference was measured midway between the iliac crest and the costal margin following a quiet expiration, and lastly hip circumference was measured at the maximal circumference over the buttocks and below the iliac crest.
blood pressure | 3 month
  Systolic and diastolic blood pressure were measured by fully automatic clinically validated blood pressure monitors (UA 779, UA-767 Plus 30 or UA 767 PC, A&D Company Ltd, Tokyo, Japan)
Aerobic fitness | after 3 month
  Estimated during a max (watt-max) or a sub-maximal test on a ergometer bike depending on the physical condition of the participant (Ergomedic 828E, Monark Exercise AB, Vansbro, Sweden). One of the following conditions contraindicated participation in the watt-max test: Any heart-related disease, chest pain, hypertension (>160/100 mmHg), heart or lung (pulmonary) medication, pregnancy and muscle, joint or skeletal problems. The sub-max test was contradicted by hypertension (>180/110 mmHg), severe heart-related disease, certain types of heart medication, muscle, joint or skeletal problems.
Arm muscle strength | after 3 month
  Arm mucle strength was measured by bending of the arms with a Takei TKK 5402 digital back strength dynamometer (Takei Scientific Instruments Co. Ltd., Tokyo, Japan). The test was performed with maximal exertion.
blood samples | After 3 months
  Non-fasting venous blood samples were collected for future analyses of P-cholesterol, P-triglyceride, and haemoglobin A1c and for biobank storage.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Wolff Hansen, Msc., Principal Investigator — National Institute of public Health
Locations (4):
- Denmark (4):
  - National Institute of Public Health, Copenhagen
  - Municipality of Frederiksberg, Frederiksberg
  - Municipality of Silkeborg, Silkeborg
  - Municipality of Varde, Varde

REFERENCES:
- [Derived] Hansen AW, Gronbaek M, Helge JW, Severin M, Curtis T, Tolstrup JS. Effect of a Web-based intervention to promote physical activity and improve health among physically inactive adults: a population-based randomized controlled trial. J Med Internet Res. 2012 Oct 30;14(5):e145. doi: 10.2196/jmir.2109. PMID 23111127